CLINICAL TRIAL: NCT03518502
Title: Comparison of Efficacy Between Sorafenib Monotherapy vs. Transarterial Chemoembolization -Sorafenib Sequential Therapy in Hepatocellular Carcinoma Patients With Extrahepatic Metastasis
Brief Title: Sorafenib Monotherapy vs. TACE-sorafenib Sequential Therapy for HCC With Metastasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University (Other)
Collaborators: Korean Liver Cancer Study Group (Other)
Responsible Party: Principal Investigator, Hyung Joon Yim, Professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012AS0313
Record Dates: First submitted 2018-04-21; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Hepatocellular Carcinoma; Metastasis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis | interventions — Sorafenib

STUDY DESIGN:
Intervention Model Description: Sorafenib monotherapy vs. transarterial chemoembolization-sorafenib sequential therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sorafenib monotherapy arm (Active Comparator): The sorafenib monotherapy group receives sorafenib immediately after randomization.
  Interventions: Drug: Sorafenib
- TACE-sorafenib sequential therapy arm (Experimental): TACE(transarterial chemoembolization )-sorafenib group receives 2~4 times of TACE before starting sorafenib.
  Interventions: Procedure: transarterial chemoembolization (TACE); Drug: Sorafenib

INTERVENTIONS:
Procedure: transarterial chemoembolization (TACE) — Standard therapy for intermediate HCC, but nor for advanced HCC
  Arms: TACE-sorafenib sequential therapy arm
Drug: Sorafenib — Standard therapy for advanced HCC

SUMMARY:
Sorafenib is the standard therapy for hepatocellular carcinoma (HCC) with extrahepatic metastasis (EHM). However, addition of transarterial chemoembolization (TACE) may be beneficial for controlling intrahepatic tumour. The investigators aimed to compare the efficacy between the sorafenib monotherapy and TACE-sorafenib sequential therapy in HCC patients with EHM.

DETAILED DESCRIPTION:
Sorafenib is the standard therapy for hepatocellular carcinoma (HCC) with extrahepatic metastasis (EHM). However, transarterial chemoembolization (TACE) which is a standard therapy for intermediate stage may be beneficial for controlling intrahepatic tumour, thereby providing chance of improving survival in HCC patients with EHM.

The investigators aimed to compare the efficacy between the sorafenib monotherapy and TACE-sorafenib sequential therapy in HCC patients with EHM.

This study is a prospective randomized controlled study being conducted at 6 tertiary hospitals in South Korea. HCC patients with EHM are being enrolled and randomized into sorafenib monotherapy or TACE-sorafenib sequential therapy group. Patients with main portal vein invasion, Child-Pugh class B or C, and history of TACE or previous systemic therapy are being excluded. The sorafenib monotherapy group receives sorafenib immediately after randomization while the TACE-sorafenib group receives 2~4 times of TACE before starting sorafenib. Response evaluation are performed every 2 months, and time to progression (TTP), progression free survival (PFS), median survival time (MST), and overall survival (OS) which is the primary outcome measure will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatocellular carcinoma by the European Association for the Study of the Liver (EASL) criteria or pathology
* One or more extrahepatic metastatic lesion by proven radiologically or histologically
* No serious coagulation abnormalities
* Performance status 0 or 1 by Eastern Cooperative Oncology Group(ECOG) criteria
* Child-Pugh score 5 or 6
* Serum creatinine <1.5mg/dL
* Age between 18 ~ 75 years old
* No other life-threatening medical illness

Exclusion Criteria:

* Patients with main portal vein invasion
* Child-Pugh class B or C
* History of TACE or previous systemic chemotherapy including sorafenib
* Age >75 years old
* Cardiovascular diseases
* History of gastrointestinal bleeding within 2 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-03-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to Feb 28, 2020 (maxium duration: up to 8 years)
  Survival rate during the study period

SECONDARY OUTCOMES:
Time to progression (TTP) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to Feb 28, 2020 (maxium duration: up to 8 years)
  Time form the enrollment to the event of progression
Progression free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to Feb 28, 2020 (maxium duration: up to 8 years)
  Survival rate without progression of HCC
Median survival time (MST) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to Feb 28, 2020 (maxium duration: up to 8 years)
  Median time of the patient survival

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Joon Yim, M.D., Principal Investigator — Korea University Ansan Hospital
Locations (6):
- South Korea (6):
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Soonchunghyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Keimyung University Dongsan Hospital, Daegu
  - Chonnam National University Hwasoon Hospital, Gwangju
  - Seoul Saint Marry Hospital, the Catholic University of Korea, Seoul
  - Severance Hospital, Yonsei University, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Result] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Result] Camma C, Schepis F, Orlando A, Albanese M, Shahied L, Trevisani F, Andreone P, Craxi A, Cottone M. Transarterial chemoembolization for unresectable hepatocellular carcinoma: meta-analysis of randomized controlled trials. Radiology. 2002 Jul;224(1):47-54. doi: 10.1148/radiol.2241011262. PMID 12091661
- [Result] Llovet JM, Bruix J. Systematic review of randomized trials for unresectable hepatocellular carcinoma: Chemoembolization improves survival. Hepatology. 2003 Feb;37(2):429-42. doi: 10.1053/jhep.2003.50047. PMID 12540794
- [Result] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Result] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Result] Cabrera R, Pannu DS, Caridi J, Firpi RJ, Soldevila-Pico C, Morelli G, Clark V, Suman A, George TJ Jr, Nelson DR. The combination of sorafenib with transarterial chemoembolisation for hepatocellular carcinoma. Aliment Pharmacol Ther. 2011 Jul;34(2):205-13. doi: 10.1111/j.1365-2036.2011.04697.x. Epub 2011 May 23. PMID 21605146